CLINICAL TRIAL: NCT04326400
Title: Active Monitoring And Determinants of Incidence Infection of COVDI-19 in a Hospital Population (AMADIICH) Study Protocol
Brief Title: Active Monitoring And Determinants of Incidence Infection of COVDI-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundación Teófilo Hernando, Spain (Other)
Responsible Party: Sponsor
Other Study IDs: AMADIICH
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Coronavirus Infection
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hospital de la Princesa employees

SUMMARY:
7. Objectives To apply e-health methods to perform active monitoring and assess determinants of incident Infection of COVID-19 in a hospital population.

8. Study design Prospective, Single-centre, observational clinical study. 9. Disease or disorder under study Healthy people in risk of COVID-19 infection. 10. Main variable. Symptoms related to infection caused by SARS-Cov2. 11. Study population and total number of patients Men and women in general god health status aged between 18 and 80 years that currently are employees of Hospital de La Princesa .

12. Duration of treatment Each subject will be monitored, since its recruitment, for a period of 12 weeks.

13. Timetable and expected date of completion The overall duration of the study is estimated at about 6 months, from patient recruitment to the last data recorded by last subject. The aim is to carry out this study from March 2020 onwards.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject age ≥ 18 years.
2. The subject has no symptoms in last week of COVID-19 infection such as:

   * Body temperature ≤ 37, 1 ºC.
   * Normal lung and breath functions.
3. The subject belongs to the Hospital de La Princesa workforce.

Exclusion Criteria:

1. People with any symptom suspicious of COVID-19 infection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in the maximum number of subjects willing to participate and able to understand and sign the informed consent form.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-03-23 (Actual); Primary Completion 2020-07-20 (Estimated); Study Completion 2020-09-20 (Estimated)

PRIMARY OUTCOMES:
COVID-19 App-based platform | 6 months
  The primary objective of this trial is to investigate whether the use of a cell phone App-based platform is a useful tool to monitor the symptoms of a population in risk of SARS-Cov2 infection. The final aim is to assess determinants of incidence of infection of COVID-19 in people working in Hospital during the pandemia of SARS-Cov-2.

SECONDARY OUTCOMES:
COVID-19 infection | 6 months
  To monitor in real-time COVID-19 symptoms in the hospital workforce, which are a proxy of incident infection (Step 1) To identify in real-time clusters of COVID-19 symptoms and to facilitate control measures.
  To determine the incidence of new infection of COVID-19. To identify the determinants and risk/protective factors associated with this infection, in a workforce hospital population free of COVID-19 at the start of our study.

CONTACTS AND LOCATIONS:
Overall Officials: Joan Soriano, MD, PhD, Principal Investigator — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Locations (1):
- Hospital Universitario de la Princesa, Madrid, Spain

REFERENCES:
- [Derived] Soriano JB, Fernandez E, de Astorza A, Perez de Llano LA, Fernandez-Villar A, Carnicer-Pont D, Alcazar-Navarrete B, Garcia A, Morales A, Lobo M, Maroto M, Ferreras E, Soriano C, Del Rio-Bermudez C, Vega-Piris L, Basagana X, Muncunill J, Cosio BG, Lumbreras S, Catalina C, Alzaga JM, Gomez Quilon D, Valdivia CA, de Lara C, Ancochea J. Hospital Epidemics Tracker (HEpiTracker): Description and pilot study of a mobile app to track COVID-19 in hospital workers. JMIR Public Health Surveill. 2020 Sep 21;6(3):e21653. doi: 10.2196/21653. PMID 32845852